CLINICAL TRIAL: NCT04270552
Title: The Effect Of Polivalent Mechanical Bacterial Lysate On The Clinical Course Of Grass Pollen-Induced Allergic Rhinitis In Children
Brief Title: Efficacy Of Bacterial Lysate In Children With Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Kamil Janeczek, MD, PhD, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KE-0254/41/2018
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; seasonal allergic rhinitis; children; grass pollen season; bacterial lysate; Th2 inflammation; eosinophils; specific immunoglobulin E
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Broncho-Vaxom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ismigen (Experimental): Treatment over 3 successive months with one daily tablet over 10 days followed by 20 days of rest.
  Interventions: Drug: Ismigen
- Placebo (Placebo Comparator): Treatment over 3 successive months with one daily tablet over 10 days followed by 20 days of rest.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ismigen — Sublingual tablets containing 7 mg of bacterial lysate from the following bacteria: Staphylococcus aureus, Haemophilus influenzae serotype B, Klebsiella pneumoniae, Klebsiella ozaenae, Neiserria catarrhalis, Streptococcus viridans, Streptococcus pyogenes, Streptococcus pneumoniae (6 strains: TY1/EQ11, TY2/EQ22, TY3/EQ14, TY5/EQ15, TY8/EQ23, TY47/EQ24) - sublingual use 1 tablet per day over 10 days for 3 successive months.
  Other Names: Polyvalent Mechanical Bacterial Lysate (PMBL)
  Arms: Ismigen
Drug: Placebo — Matched tablets without any active substance.
  Arms: Placebo

SUMMARY:
This study evaluate the efficacy of Polyvalent Mechanical Bacterial Lysate (PMBL - Ismigen) to improve the clinical course of grass pollen-induced allergic rhinitis (using: TNSS, TOSS, VAS, PNIF) in children aged 5 to 17. Half of the 70 participants will receive PMBL while the other half will receive placebo.

DETAILED DESCRIPTION:
Seasonal allergic rhinitis (SAR) is caused by the allergens of wind-pollinated plants, and in Poland mainly by grass pollen allergens. During the grass pollen season, patients may suffer from fatigue, weakness, lack of fitness, difficulty in sleeping and reduced performance at school. In people allergic to the above-mentioned pollen, the disease significantly reduces the quality of life and requires intensive treatment in the pollen period.

Due to the high incidence of allergic rhinitis, the negative impact of the disease on the quality of life, and incomplete effectiveness of previously available therapeutic methods, new methods of treatment are being developed. Recent research highlights the immunoregulatory potential of bacterial lysates, indicating the possibility of their future use in the prevention and treatment of allergic diseases, including atopic dermatitis, allergic rhinitis, and asthma. However, so far no randomized, double-blind, placebo-controlled, study with bacterial lysate in children's SAR therapy has been conducted.

The main aim of this study was to evaluate the clinical course of the pollen allergic rhinitis, caused by grass pollen allergens in children during the grass pollen season, treated with polyvalent mechanical bacterial lysate (PMBL). The approval of the Bioethics Committee at the Medical University in Lublin was obtained for the study.

Seventy children with SAR were enrolled to this study and were randomly assigned to the PMBL group (n=35) and placebo group (n=35). Three visits took place as part of the study: at the beginning of the grass pollen season, at the peak, and at the end of the season. The time frame of the grass pollen season for south-eastern Poland was determined using the "95%" method on the basis of measurements of grass pollen concentration in the atmospheric air, which were obtained from the Environmental Allergy Research Centre in Warsaw.

Nasal and ocular SAR symptoms were recorded by parents of children in the daily patient diary according to the standard scoring systems (TNSS, total nasal symptom score and TOSS, total ocular symptom score), and their intensity was also evaluated during three visits using VAS (visual analogue scale). At each visit, peak nasal inspiratory flow (PNIF) was also measured.

In order to determine the mechanism responsible for the possible effects of PMBL, samples were taken from patients for additional testing: nasal smears for the presence of eosinophils and nasal lavage fluids for the presence of allergen-specific IgE (asIgE) against timothy grass pollen allergens.

ELIGIBILITY:
Inclusion Criteria:

1. Children of both genders aged 5 to 17 years.
2. Children with grass pollen-induced allergic rhinitis recognized and treated according to current ARIA (Allergic Rhinitis and its Impact on Asthma) recommendations.
3. Positive skin prick test to grass pollen allergens or positive specific IgE (defined as ≥ class 2, ≥ 0,70 kU/l) against timothy grass pollen allergens.
4. Presentation of clinical symptoms of the allergic rhinitis (rhinorrhea, nasal congestion, nasal itching, sneezing) in at least two recent grass pollen seasons in Poland before inclusion in the study.
5. Proper use of PMBL sublingual tablets.
6. Written informed consent obtained from parents/guardians before any study related procedures are performed.

Exclusion Criteria:

1. Patient received mechanical or any other polyvalent bacterial lysate immunostimulation within the previous 12 months before visit 1.
2. Patient received oral/subcutaneous allergen-immunotherapy within the previous 3 years before the start of the study.
3. Vaccination performed within 3 months before the beginning of the study.
4. Deficiencies in cellular and humoral immunity.
5. Treatment with systemic corticosteroids within the last 6 months before the start of the study.
6. Pregnant or breastfeeding woman.
7. Other chronic conditions of the nose or nasal sinuses.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2018-04-22 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-12 (Actual)

PRIMARY OUTCOMES:
Change in the severity of nasal SAR symptoms as assessed by Total Nasal Symptom Score (TNSS) | at baseline, at 1-month, at 2-months and at 3-months
  The severity of nasal SAR symptoms (sneezing, runny nose, itchy nose and nasal congestion) were recorded by parents of children in the daily patient diary using the following scale: 0 = absent (no symptom); 1 = mild (symptom present, easily tolerated); 2 = moderate (awareness of symptom, bothersome but tolerable); 3 = severe (symptoms hard to tolerate, interfere with daily activities and/or sleeping).
  The Total Nasal Symptom Score (sum of the 4 symptom scores) ranges from 0 (no symptoms) to 12 (worst symptoms).
  Weekly average TNSS values from the baseline period (beginning of the grass pollen season) and obtained 1 month (grass pollen season - significant intensification of SAR symptoms), 2 months (peak grass pollen season) and 3 months (3 weeks before the end of the grass pollen season) after initiating therapy were used for statistical analysis.
Change in the severity of ocular SAR symptoms as assessed by Total Ocular Symptom Score (TOSS) | at baseline, at 1-month, at 2-months and at 3-months
  The severity of ocular SAR symptoms (redness of the eyes, watery eyes, itching of the eyes) were recorded by parents of children in the daily patient diary using the following scale: 0 = absent (no symptom); 1 = mild (symptom present, easily tolerated); 2 = moderate (awareness of symptom, bothersome but tolerable); 3 = severe (symptoms hard to tolerate, interfere with daily activities and/or sleeping).
  The Total Ocular Symptom Score (sum of the 3 symptom scores) ranges from 0 (no symptoms) to 9 (worst symptoms).
  Weekly average TOSS values from the baseline period (beginning of the grass pollen season) and obtained 1 month (grass pollen season - significant intensification of SAR symptoms), 2 months (peak grass pollen season) and 3 months (3 weeks before the end of the grass pollen season) after initiating therapy were used for statistical analysis.
Change in the nasal obstruction using Peak Nasal Inspiratory Flow (PNIF) | at baseline, at 2-months and at 3-months
  Assessment of the nasal obstruction before (visit 1) and 2 months (visit 2) and 3 months (visit 3) after initiating therapy based on measurement of Peak Nasal Inspiratory Flow by Youlten Peak Flow Meter (Clement Clarke International, UK).
  The higher PNIF value, the smaller nasal obstruction.
Change in the severity of nasal SAR symptoms as assessed by Visual Analogue Scale (VAS) | at baseline, at 2-months and at 3-months
  Assessment of the severity of nasal SAR symptoms before (visit 1) and 2 months (visit 2) and 3 months (visit 3) after initiating therapy with the use of Visual Analogue Scale.The patient was asked to indicate the severity of nasal SAR symptoms on a 100 mm Visual Analogue Scale, were 0 is no symptoms and 100 the worst possible symptoms.
Change in the severity of ocular SAR symptoms as assessed by Visual Analogue Scale (VAS) | at baseline, at 2-months and at 3-months
  Assessment of the severity of ocular SAR symptoms before (visit 1) and 2 months (visit 2) and 3 months (visit 3) after initiating therapy with the use of Visual Analogue Scale. The patient was asked to indicate the severity of ocular SAR symptoms on a 100 mm Visual Analogue Scale, were 0 is no symptoms and 100 the worst possible symptoms.

SECONDARY OUTCOMES:
Nasal eosinophil count | at baseline, at 2-months and at 3-months
  To assess the change in the number of eosinophils in nasal smears.
Specific immunoglobulin E concentration | at baseline, at 2-months and at 3-months
  To assess the change in the level of allergen-specific immunoglobulin E (asIgE) against timothy grass pollen allergens in nasal lavage fluid and blood serum.
Frequency of oral H1-antihistamines use | from baseline, up to the 3-month time point
  To assess the mean number of days of oral H1-antihistamines use for the relief of SAR symptoms.
Frequency of intranasal corticosteroids use | from baseline, up to the 3-month time point
  To assess the mean number of days of intranasal corticosteroids use for the relief of SAR symptoms.
Incidence of treatment emergent adverse events [safety and tolerability] | from baseline, up to the 3-month time point
  Incidence, frequency and severity of treatment emergent adverse events.
Incidence of treatment emergent adverse events leading to discontinuation [safety and tolerability] | from baseline, up to the 3-month time point
  The number of participants with adverse events leading to discontinuation.
Time to discontinuation due to treatment emergent adverse events [safety and tolerability] | From date of randomization until the date of occurrence of an adverse event leading to discontinuation, assessed up to 3 months
  To assess the time that has elapsed since treatment initiation to the occurrence of an adverse event leading to discontinuation.
Incidence of treatment emergent clinical laboratory test abnormalities [safety and tolerability] | at baseline and at 3-months
  Complete blood count assessment at baseline and at 3-months.
Incidence of treatment emergent abnormalities in physical examination findings [safety and tolerability] | at baseline, at 2-months and at 3-months
  Observe skin, lymph nodes, ears, eyes, nose, throat, cardiac and pulmonary status, abdomen and extremities for any abnormalities.
Incidence of treatment emergent abnormalities in pulse rate [safety and tolerability] | at baseline, at 2-months and at 3-months
  Measure resting pulse rate as beats per minute.
Incidence of treatment emergent abnormalities in blood pressure [safety and tolerability] | at baseline, at 2-months and at 3-months
  Measure systolic and diastolic blood pressure (in mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary Diseases and Children Rheumatology, Medical University of Lublin, Lublin, Poland

REFERENCES:
- [Background] Janeczek KP, Emeryk A, Rapiejko P. Effect of polyvalent bacterial lysate on the clinical course of pollen allergic rhinitis in children. Postepy Dermatol Alergol. 2019 Aug;36(4):504-505. doi: 10.5114/ada.2019.87457. Epub 2019 Aug 30. No abstract available. PMID 31616231
- [Background] Banche G, Allizond V, Mandras N, Garzaro M, Cavallo GP, Baldi C, Scutera S, Musso T, Roana J, Tullio V, Carlone NA, Cuffini AM. Improvement of clinical response in allergic rhinitis patients treated with an oral immunostimulating bacterial lysate: in vivo immunological effects. Int J Immunopathol Pharmacol. 2007 Jan-Mar;20(1):129-38. doi: 10.1177/039463200702000115. PMID 17346436
- [Background] Meng Q, Li P, Li Y, Chen J, Wang L, He L, Xie J, Gao X. Broncho-vaxom alleviates persistent allergic rhinitis in patients by improving Th1/Th2 cytokine balance of nasal mucosa. Rhinology. 2019 Dec 1;57(6):451-459. doi: 10.4193/Rhin19.161. PMID 31403136
- [Background] Han L, Zheng CP, Sun YQ, Xu G, Wen W, Fu QL. A bacterial extract of OM-85 Broncho-Vaxom prevents allergic rhinitis in mice. Am J Rhinol Allergy. 2014 Mar-Apr;28(2):110-6. doi: 10.2500/ajra.2013.27.4021. PMID 24717947
- [Background] Liu C, Huang R, Yao R, Yang A. The Immunotherapeutic Role of Bacterial Lysates in a Mouse Model of Asthma. Lung. 2017 Oct;195(5):563-569. doi: 10.1007/s00408-017-0003-8. Epub 2017 May 4. PMID 28474108
- [Background] Esposito S, Soto-Martinez ME, Feleszko W, Jones MH, Shen KL, Schaad UB. Nonspecific immunomodulators for recurrent respiratory tract infections, wheezing and asthma in children: a systematic review of mechanistic and clinical evidence. Curr Opin Allergy Clin Immunol. 2018 Jun;18(3):198-209. doi: 10.1097/ACI.0000000000000433. PMID 29561355
- [Background] Emeryk A, Bartkowiak-Emeryk M, Raus Z, Braido F, Ferlazzo G, Melioli G. Mechanical bacterial lysate administration prevents exacerbation in allergic asthmatic children-The EOLIA study. Pediatr Allergy Immunol. 2018 Jun;29(4):394-401. doi: 10.1111/pai.12894. PMID 29575037
- [Result] Janeczek K, Emeryk A, Rachel M, Duma D, Zimmer L, Poleszak E. Polyvalent Mechanical Bacterial Lysate Administration Improves the Clinical Course of Grass Pollen-Induced Allergic Rhinitis in Children: A Randomized Controlled Trial. J Allergy Clin Immunol Pract. 2021 Jan;9(1):453-462. doi: 10.1016/j.jaip.2020.08.025. Epub 2020 Aug 26. PMID 32858239